CLINICAL TRIAL: NCT06335966
Title: Barrett's Esophagus Screening Towards Rural Referral Pathways: Screening for Esophageal Cancer in Rural Oregon Without Endoscopy
Brief Title: BEST-RPP Pilot: Screening for Esophageal Cancer in Rural Oregon Without an Endoscopy
Acronym: BEST-RPP
Status: Active, not recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Kuni Foundation (Unknown); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Fouad Otaki, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00025975
Record Dates: First submitted 2024-02-08; First posted 2024-03-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with suspected Barrett's Esophagus or at risk for esophageal cancer: Patients who receive primary care in a rural settings and are in need of screening for Barrett's Esophagus or esophageal cancer.
  Interventions: Device: Screening with swallowable esophageal cell-collection devices (SECD)

INTERVENTIONS:
Device: Screening with swallowable esophageal cell-collection devices (SECD) — All participants who enroll in this study and provide their consent will undergo screening with an FDA approved swallowable esophageal cell-collection device (SECD)

SUMMARY:
Recent advancements in swallowable esophageal cell-collection devices (SECD) offer a safe, minimally invasive, accurate, and low-cost alternative to esophageal screening without the need for an upper endoscopy. The BEST-RPP study aims to evaluate the acceptability and feasibility of using this novel approach to screen for Barrett's Esophagus (BE) and Esophageal Carcinoma (EAC) in rural primary care clinic settings in Oregon.

DETAILED DESCRIPTION:
This is a proof-of-concept observational study to pilot the use of an FDA approved swallowable esophageal cell-collection device to screen for esophageal cancer in two rural primary care clinics in Oregon. The principal investigator will work with clinic staff to gauge the current use and understanding of SECDs as screening tools for esophageal cancer and to identify 50 patients at each site to approach about SECDs as an option for screening, for a total of 100 patients. If patients provide their consent and are eligible, they will undergo SECD administration for cancer screening in their primary care clinic. The study will evaluate the feasibility of use of this diagnostic tool in rural primary care settings, patient acceptability of screening for esophageal cancer via SECD in their primary care clinics, and where there are positive cases, the efficacy of diagnostic and treatment pathways to transitioning patients to tertiary centers for full diagnostic workup.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Willing and able to comply with the protocol
* Live in a rural area
* Chronic GERD Dx
* 3 or more of the following risk factors: Male, age >50 years White race Tobacco smoking Obesity Family history of BE or EAC in a first-degree relative

Exclusion Criteria:

-

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study seeks to enroll patients who: live in a rural area as defined by a Rural-Urban Commuting Area Code (RUCA) of greater than 4, are ages 50 years and above, and have screening as indicated by the American College of Gastroenterology recommendations for EAC (list below).
  * Chronic GERD Dx
  * 3 or more risk factors:
    * Male, age >50 years
    * White race
    * Tobacco smoking
    * Obesity
    * Family history of BE or EAC in a first-degree relative
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the use of a SECD: Number of providers who indicate likelihood of using SECD | 8 months
  Feasibility of screening for esophageal cancer via SECD in rural primary care settings will be measured by data collected from Provider Post-Inservice Questionnaire, which includes, Indication of provider likelihood of using SECD as a screening tool.
Feasibility of the use of SECD: Number of providers who indicate willingness to be trained and train clinic staff | 8 months
  Feasibility of screening for esophageal cancer via SECD in rural primary care settings will be measured by data collected from Provider Post-Inservice Questionnaire, which includes, Indication of provider willingness to be trained and train clinic staff in SECD administration.
Feasibility of the use of SECD: Number of referrals | 8 months
  Feasibility of screening for esophageal cancer via SECD in rural primary care settings will be measured by data collected from number of provider referrals received for the study.
Feasibility of the use of SECD: Number enrolled | 8 months
  Feasibility of screening for esophageal cancer via SECD in rural primary care settings will be measured by data collected from number of patients enrolled.
Patient acceptability: Number of interested patients who schedule an appointment to be screened | 8 months
  Assess patient acceptability of using a SECD for screening in rural primary care settings vs tertiary care centers Acceptability will be measured by the number of interested patients who schedule an appointment to be screened via the SECD and the number of patients who come to their appointments. As well as patients who are interested in being screened via SECD at other care centers where it is offered.
Patient acceptability: Number of patients who come to their appointments | 8 months
  Assess patient acceptability of using a SECD for screening in rural primary care settings vs tertiary care centers Acceptability will be measured by the number of interested patients who schedule an appointment to be screened via the SECD and the number of patients who come to their appointments. As well as patients who are interested in being screened via SECD at other care centers where it is offered.
Patient acceptability: Number of patients interested in being screened via SECD at other care centers | 8 months
  Assess patient acceptability of using a SECD for screening in rural primary care settings vs tertiary care centers Acceptability will be measured by the number of interested patients who schedule an appointment to be screened via the SECD and the number of patients who come to their appointments. As well as patients who are interested in being screened via SECD at other care centers where it is offered.

SECONDARY OUTCOMES:
Access: time to full diagnostic work up for patients with positive SECD results | 8 months
  Observe the time, effort, and barriers patients who live in rural areas with positive SECD tests experience to complete standard - diagnostic work up at tertiary care centers

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States